CLINICAL TRIAL: NCT02788721
Title: Assessment of Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Oral Doses of GLPG2451 and of the Combination of GLPG2451 and GLPG2222 in Healthy Female Subjects
Brief Title: A Study to Assess Safety, Tolerability and Pharmacokinetics of GLPG2451 in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Collaborators: Pharmaceutical Research Associates (Other); SGS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG2451-CL-101
Record Dates: First submitted 2016-05-13; First posted 2016-06-02 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLPG2451 single dose (Experimental): Single dose of GLPG2451 oral suspension at up to 4 dose levels in ascending order
  Interventions: Drug: GLPG2451 single dose
- Placebo single dose (Placebo Comparator): Single dose of Placebo oral suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG2451 single dose — GLPG2451 oral suspension, single ascending doses, daily
  Arms: GLPG2451 single dose
Drug: Placebo — Placebo, oral suspension, daily
  Arms: Placebo single dose

SUMMARY:
The study is a First-in-Human, Phase I, randomized, double-blind, placebo-controlled study evaluating single and multiple ascending oral doses of GLPG2451 and combined multiple doses of GLPG2451 and GLPG2222 in healthy female subjects. The purpose of the study is to evaluate safety and tolerability after single ascending oral doses and of multiple doses of GLPG2451 given to healthy female subjects compared to placebo as well as of multiple doses of the combination of GLPG2451/GLPG2222 compared to GLPG2451/placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18-65 years of age inclusive, on the day of signing informed consent form (ICF).
* Of non-childbearing potential defined as surgically sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy), or post-menopausal (at least 12 consecutive months without menstruation, without an alternative medical cause [including hormone replacement therapy]). In addition a determination of follicle stimulating hormone (FSH) can be performed with FSH >35 mIU/ml to further confirm postmenopausal status without menstruation for ≥12 months.
* A body mass index (BMI) between 18-30 kg/m2, inclusive.
* Judged by the investigator to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), Holter monitoring and a laboratory profile prior to the initial study drug administration.
* Discontinuation of all medications (including over-the-counter medications and herbal supplements) except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks) at least 2 weeks prior to the first study drug administration. In addition, subjects must agree not to take any medications (including over-the-counter medication and herbal supplements), or alcohol during the course of the study.-non-smokers and non-users of any nicotine-containing products.
* Non-smokers and non-users of any nicotine-containing products. A non-smoker is defined as an individual who has abstained from smoking for at least 1 year prior to the screening. A non-user is defined as an individual who has abstained from any nicotine containing products for at least 1 year prior to the screening.
* Negative urine drug screen (amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, and tricyclic antidepressants) and alcohol breath test.
* Able and willing to sign the ICF as approved by the IEC, prior to screening evaluations, and willing to adhere to the prohibitions and restrictions.

Exclusion Criteria:

* Known hypersensitivity or a significant allergic reaction to any drug as determined by the investigator, such as anaphylaxis requiring hospitalization.
* Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or any history of hepatitis from any cause with the exception of hepatitis A.
* History of or a current immunosuppressive condition (e.g., human immunodeficiency virus [HIV] infection).
* Symptoms of clinically significant illness in the 3 months before the initial study drug administration.
* Presence or having sequelae of gastrointestinal, liver or kidney (creatinine clearance ≤ 80 mL/min using the Cockroft formula; if calculated result ≤ 80 mL/min, a 24-hour urine collection to determine actual value can be done) or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of malignancy within the past 5 years (except for basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been treated with no evidence of recurrence).
* Clinically relevant abnormalities detected on ECG and/or Holter regarding either rhythm or conduction (e.g. QTcF ≥ 470 msec, or a known long QT syndrome). A first degree heart block will not be considered as a significant abnormality.
* Family history (if known) of long QT syndrome in a primary relative.
* Clinically relevant abnormalities detected on vital signs.
* Significant blood loss (including blood donation [> 500 mL]), or having had a transfusion of any blood product within 12 weeks prior to the initial study drug administration.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Change versus placebo in the proportion of subjects with adverse events | Between screening and 182 days after the last dose
  To assess safety and tolerability of single ascending doses with GLPG2451 versus placebo in healthy subjects

SECONDARY OUTCOMES:
Maximum observed plasma concentration of GLPG2451 (Cmax) given alone | Between day 1 predose and 175 days after the last dose
  To characterize pharmacokinetics of GLPG2451 and its metabolite after a single oral dose in healthy subjects
Time of occurrence of Cmax for GLPG2451 and (tmax) given alone | Between day 1 predose and 175 days after the last dose
  To characterize pharmacokinetics of GLPG2451 and its metabolite after a single oral dose in healthy subjects
Area under the plasma concentration-time curve (AUC0-t) of GLPG2451 given alone | Between day 1 predose and 175 days after the last dose
  To characterize pharmacokinetics of GLPG2451 and its metabolite after a single oral dose in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Chris Brearley, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided